CLINICAL TRIAL: NCT03050450
Title: A Phase 1 Study of Lenalidomide in Combination With Vorinostat in Pediatric Patients With High Grade or Progressive Central Nervous System Tumors
Brief Title: Study of Lenalidomide With Vorinostat in Pediatric Patients With High Grade or Progressive CNS Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of feasibility to accrue patients in allotted time.
Sponsor: Johns Hopkins All Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACH-CNS-005
Record Dates: First submitted 2016-08-30; First posted 2017-02-13 (Actual); Results first posted 2021-04-05 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-03

CONDITIONS: Central Nervous System Tumors
MeSH Terms: conditions — Central Nervous System Neoplasms | interventions — Lenalidomide; Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- dose level 1 (Experimental): 25 mg/m2 Lenalidomide (Revlimid®) and 180 mg/m2 Vorinostat (Zolinza®)
  Interventions: Drug: 25 mg/m2 Lenalidomide (Revlimid®) and 180 mg/m2 Vorinostat (Zolinza®)
- dose level 2 (Experimental): 50 mg/m2 Lenalidomide (Revlimid®) and 180 mg/m2 Vorinostat (Zolinza®)
  Interventions: Drug: 50 mg/m2 Lenalidomide (Revlimid®) and 180 mg/m2 Vorinostat (Zolinza®)
- dose level 3 (Experimental): 100 mg/m2 Lenalidomide (Revlimid®) and 180 mg/m2 Vorinostat (Zolinza®)
  Interventions: Drug: 100 mg/m2 Lenalidomide (Revlimid®) and 180 mg/m2 Vorinostat (Zolinza®)
- dose level 4 (Experimental): 150 mg/m2 Lenalidomide (Revlimid®) and 180 mg/m2 Vorinostat (Zolinza®)
  Interventions: Drug: 150 mg/m2 Lenalidomide (Revlimid®) and 180 mg/m2 Vorinostat (Zolinza®)
- dose level 5 (Experimental): 150 mg/m2 Lenalidomide (Revlimid®) and 230 mg/m2 Vorinostat (Zolinza®)
  Interventions: Drug: 150 mg/m2 Lenalidomide (Revlimid®) and 230 mg/m2 Vorinostat (Zolinza®)

INTERVENTIONS:
Drug: 25 mg/m2 Lenalidomide (Revlimid®) and 180 mg/m2 Vorinostat (Zolinza®) — Drug: Lenalidomide 25 mg/m2 days 1-21 of a 28 days cycle Drug: Vorinostat 180 mg/m2 days 1-7 and 15-21 of a 28 day cycle
  Other Names: Revlimid®; Zolinza®
  Arms: dose level 1
Drug: 50 mg/m2 Lenalidomide (Revlimid®) and 180 mg/m2 Vorinostat (Zolinza®) — Drug: Lenalidomide 50 mg/m2 days 1-21 of a 28 days cycle Drug: Vorinostat 180 mg/m2 days 1-7 and 15-21 of a 28 day cycle
  Other Names: Revlimid®; Zolinza®
  Arms: dose level 2
Drug: 100 mg/m2 Lenalidomide (Revlimid®) and 180 mg/m2 Vorinostat (Zolinza®) — Drug: Lenalidomide 100 mg/m2 days 1-21 of a 28 days cycle Drug: Vorinostat 180 mg/m2 days 1-7 and 15-21 of a 28 day cycle
  Other Names: Revlimid®; Zolinza®
  Arms: dose level 3
Drug: 150 mg/m2 Lenalidomide (Revlimid®) and 180 mg/m2 Vorinostat (Zolinza®) — Drug: Lenalidomide 150 mg/m2 days 1-21 of a 28 days cycle Drug: Vorinostat 180 mg/m2 days 1-7 and 15-21 of a 28 day cycle
  Other Names: Revlimid®; Zolinza®
  Arms: dose level 4
Drug: 150 mg/m2 Lenalidomide (Revlimid®) and 230 mg/m2 Vorinostat (Zolinza®) — Drug: Lenalidomide 150 mg/m2 days 1-21 of a 28 days cycle Drug: Vorinostat 230 mg/m2 days 1-7 and 15-21 of a 28 day cycle
  Other Names: Revlimid®; Zolinza®
  Arms: dose level 5

SUMMARY:
Independently, both lenalidomide and vorinostat have shown promising activity in pediatric central nervous system (CNS) tumors. These are both agents that are not typically part of first-line studies, although both agents are of serious interest and are currently in clinical trials for further investigation. This study is to evaluate the combination of lenalidomide and vorinostat in high grade or progressive central nervous system tumors in children.

DETAILED DESCRIPTION:
Brain tumors are the second most common cause of cancer in pediatrics and the leading cause of cancer death in children. For children with relapsed, refractory, or recurrent brain tumors, new agents in new combinations are needed. This study is a phase I study designed to provide an objective observation of toxicity and establish a maximum tolerated dose of this combination. In addition, this study will observe the response of children with relapsed or refractory central nervous system tumors. Lenalidomide will be dosed orally once daily days 1-21 consecutive days of a 28 day cycle. Vorinostat will be dosed orally once daily days 1-7 and 15-21 of a 28-day cycle.Doses will be escalated according to standard phase 1 dose escalation criteria. In the absence of treatment delays due to adverse event(s), treatment may continue for 24 cycles.

ELIGIBILITY:
Inclusion Criteria:

* Must have histologically confirmed central nervous system malignancy for which standard curative measures do not exist or are not loner effective
* Must have measurable disease
* may not have received vorinostat and lenalidomide in combination
* At least 3 weeks since prior chemotherapy
* At least 6 weeks from last nitrosurea
* At least 6 weeks from autologous transplant
* At least 3 months from bone marrow donor transplant
* At least 3 weeks from focal radiation
* At least 6 weeks from craniospinal radiation
* Must have not received growth factors within 1 week of study entry
* Must be on a stable or decreasing dose of steroids for 1 week prior
* Must not be receiving any chemo, biologic, or radiation therapy
* Must not be receiving enzyme inducing anticonvulsants or valproic acid
* Must not be receiving pro-thrombotic agents
* Karnofsky or Lansky performance status ≥50%
* Life expectancy of greater than 8 weeks
* Patients must have normal organ and marrow function, including
* Absolute neutrophil count ≥1,000/mcL
* Platelets ≥100,000/mcL
* Pulse oximetry >93%
* Total bilirubin ≤ 1.5 x upper limit of normal (ULN)
* aspartate aminotransferase (AST)(SGOT)/Alanine transaminase (ALT)(SGPT) ≤2.5 × institutional upper limit of normal
* Creatinine within normal institutional limits OR
* Creatinine clearance ≥60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
* The effects of vorinostat and lenalidomide on the developing human fetus are unknown. For this reason and because agents used in this trial are known to be teratogenic, women of child-bearing potential must commit to complete abstinence or use TWO methods of birth control (one highly effective (i.e. intrauterine device (IUD), birth control pills, injections, implants, tubal ligation, partner's vasectomy), and one additional method (i.e. male condom, diaphragm, cervical cap) for the duration of study participation and at least 28 days after completion. Females of childbearing potential must agree to ongoing pregnancy testing and counseling every 28 days about pregnancy precautions. If a female has not had a menstrual period in the preceding 24 consecutive months or has had a hysterectomy, the two methods of birth control requirement does not apply. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must agree to use condoms for the duration of study participation, and 28 days after completion.

Exclusion Criteria:

* Patient has not recovered from acute toxic effects of all prior therapies
* Patients who are receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to vorinostat or lenalidomide
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, dyspnea at rest, symptomatic congestive heart failure, history of thromboembolism unrelated to central line, patients with known predisposition syndrome for thromboembolism, patients receiving anticoagulation therapy, unstable angina pectoris, cardiac arrhythmia, patients receiving enzyme inducing anticonvulsants, patients receiving valproic acid, patients receiving antiplatelet agents (aspirin, anti-inflammatory drugs), or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study due to the potential for teratogenic effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with these agents, breastfeeding should be discontinued if the mother is being treated and not resumed until 28 days after completing therapy.
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with these agents. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy.

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2016-08-10 (Actual); Primary Completion 2018-12-19 (Actual); Study Completion 2018-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stacie Stapleton, MD, Principal Investigator — Johns Hopkins All Children's Hospital
Locations (1):
- Johns Hopkins All Childen's Hospital, St. Petersburg, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 2 participants were unable to start because they couldn't swallow pills. Study did not proceed beyond dose level 1.
Period: Overall Study
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4 | Dose Level 5
Started | 6 | 0 | 0 | 0 | 0
Completed | 5 | 0 | 0 | 0 | 0
Not Completed | 1 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Did not go past dose level 1
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4 | Dose Level 5 | Total
Number analyzed (Participants) | 6 | 0 | 0 | 0 | 0 | 6
Age, Continuous [Median (Full Range); unit: years] | 7.1 [1.9 to 8.7] |  |  |  |  | 7.1 [1.9 to 8.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 |  |  |  |  | 4
  Male | 2 |  |  |  |  | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 |  |  |  |  | 1
  Not Hispanic or Latino | 5 |  |  |  |  | 5
  Unknown or Not Reported | 0 |  |  |  |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  |  |  |  | 0
  Asian | 0 |  |  |  |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  |  |  |  | 0
  Black or African American | 4 |  |  |  |  | 4
  White | 2 |  |  |  |  | 2
  More than one race | 0 |  |  |  |  | 0
  Unknown or Not Reported | 0 |  |  |  |  | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 |  |  |  |  | 6
Diagnosis [Count of Participants; unit: Participants]
  Low Grade Glioma | 1 |  |  |  |  | 1
  High Grade Glioma | 1 |  |  |  |  | 1
  ATRT | 1 |  |  |  |  | 1
  Ependymoma | 2 |  |  |  |  | 2
  DIPG | 1 |  |  |  |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Adverse Events
Description: Collect and grade all of the adverse events to evaluate for safety. This data was collected for the first 2 cycles for each participant.
Time Frame: Two 28 day cycles
Population: Did not go beyond dose level 1.
Measure: Number; unit: total adverse events
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4 | Dose Level 5
Number analyzed (Participants) | 6 | 0 | 0 | 0 | 0
total adverse events
  Grade 1 adverse events | 68 |  |  |  |
  Grace 2 adverse events | 32 |  |  |  |
  Grade 3 adverse events | 12 |  |  |  |
  Grade 4 adverse events | 2 |  |  |  |
  Grade 5 adverse events | 1 |  |  |  |

2. Secondary Outcome: Best Response of Children With Recurrent or Refractory Central Nervous System Tumors
Description: Best response by MRIs per definitions in the protocol (complete response, partial response, stable disease, progressive disease). MRI's were obtained every 2 cycles and the best response was reported.
Time Frame: Every 2 cycles up to 24 cycles
Population: Did not go beyond dose level 1. 4 participants were assessed for this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4 | Dose Level 5
Number analyzed (Participants) | 4 | 0 | 0 | 0 | 0
Participants
  Complete Response | 0 |  |  |  |
  Partial Response | 1 |  |  |  |
  Stable Disease | 1 |  |  |  |
  Progressive Disease | 2 |  |  |  |

3. Secondary Outcome: 2 Year Event Free Survival With Children Treated With This Regimen.
Description: 2 year actual event free survival with children treated with this protocol.
Time Frame: 2 year
Population: Data was not collected for this outcome measure.
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4 | Dose Level 5
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Number Participants With Hematologic and Non-hematologic Toxicities
Description: Number participants with grades 3 to 5 hematologic and non-hematologic toxicities. All toxicities are for end of cycle 2.
Time Frame: Two 28 day cycles
Population: Did not go beyond dose level 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4 | Dose Level 5
Number analyzed (Participants) | 6 | 0 | 0 | 0 | 0
Participants
  Grade 3 & 4 Blood/Bone Marrow | 0 |  |  |  |
  Grade 3 & 4 Gastrointestinal | 2 |  |  |  |
  Grade 3 & 4 Metabolic/Laboratory | 5 |  |  |  |
  Grade 3 & 4 Musculoskelatal/Soft Tissue | 1 |  |  |  |
  Grade 3 & 4 Neurology | 1 |  |  |  |
  Grade 3 & 4 Pain | 0 |  |  |  |
  Grade 3 & 4 Vascular | 0 |  |  |  |
  Grade 3 & 4 & 5 Other | 6 |  |  |  |

ADVERSE EVENTS:
Time Frame: Two 28 day cycles for each patient
Description: did not go beyond dose level 1
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4 | Dose Level 5
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 2/6 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 2/6 | 0/0 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 (N=6) | Dose Level 2 (N=0) | Dose Level 3 (N=0) | Dose Level 4 (N=0) | Dose Level 5 (N=0)
Hospitalized for ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — This Serious Adverse Event (SAE) was related to disease - the patient hospitalized for ascites and found to have peritoneal seeding via ventriculoperitoneal shunt
Hospitalized for abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Patient with G-tube hospitalized for abdominal pain and observed and discharged.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 (N=6) | Dose Level 2 (N=0) | Dose Level 3 (N=0) | Dose Level 4 (N=0) | Dose Level 5 (N=0)
Grade 3-4 (Blood and lymphatic system disorders) | 2 (3) | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-10-05): https://cdn.clinicaltrials.gov/large-docs/50/NCT03050450/SAP_000.pdf
  • Study Protocol and Informed Consent Form (2018-10-05): https://cdn.clinicaltrials.gov/large-docs/50/NCT03050450/Prot_ICF_001.pdf